CLINICAL TRIAL: NCT06447818
Title: Changes in Difficult Airway Markers After Surgery for Obstructive Sleep Apnoea Syndrome
Status: Recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-40
Record Dates: First submitted 2024-05-20; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea of Adult; Difficult or Failed Intubation
Keywords: Obstructive sleep apnea surgery, Difficult airway markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway groups: This group will consist of patients who will undergo airway surgery for obstructive sleep apnoea
  Interventions: Other: Change in airway markers

INTERVENTIONS:
Other: Change in airway markers — Mallampati and cormack lahane scores will be evaluated at the sixth postoperative month

SUMMARY:
This study investigates the changes in difficult airway markers at 6 months post operatively in patients undergoing obstructive sleep apnoea surgery

DETAILED DESCRIPTION:
The incidence of difficult airway is approximately one in 1000 cases and it is a life-threatening condition in perioperative patients. Many classifications, guidelines and appæroaches have been proposed to recognise patients with difficult airway. Even the most well-known classifications are not 100% successful in predicting difficult airway . For this reason, some unexpected difficult airway cases are encountered and their management is the subject of new research in the literature .

Obstructive sleep apnoea syndrome (OSAS) is associated with the possibility of difficult airway. Perioperative airway complications may also increase in patients with OSAS. Complications related with cardiac, pulmonary, endocrine and other systems are observed in patients living with a diagnosis of OSAS for a long time. The rate of complications is increased especially in patients with prolonged apnoea episodes during sleep.Anaesthesia process also poses a risk for OSAS patients. In patients receiving positive airway pressure therapy at home, intensive care or close anaesthesia is required at the end of the operation.follow-up is applied. In addition, OSAS patients are suitable candidates for day surgery, which is increasing day by day.

Reducing the symptoms with surgical treatment before OSAS is complicated can also reduce the effects that may occur in the future. Surgeries such as anterior uvulopalatinoplasty are frequently performed in these patients. OSAS patients require close follow-up and evaluation in terms of anaesthesia before these surgeries. A decrease in symptoms after surgery has been shown in some publications.Our study will be conducted in prospective observational status. Within the study period (01.05.2024-01.05.2025), patients who will undergo OSAS surgery by the ENT clinic in our operating theatres in a 12-month period will be included. In the preoperative evaluation of these patients; STOP-BANG and Epworth sleepiness test, SF-12 quality of life scales and laboratory values, if any, echocardiography results will be collected.

Weight, mallampati scores, neck circumference, thyromental distances and demographic data will be recorded at the preoperative visit.

After induction of anaesthesia, parameters such as mask ventilation, difficulty in laryngoscopy and intubation, Cormack-Lehane scores on direct laryngoscopy and the need for advanced airway techniques will be recorded.

At the end of the operation, the type of surgery performed and the need for intensive care will be recorded.

Patients will be routinely awakened and extubated at the end of the operation and discharged home with routine procedures after follow-up in the ward. Due to its observational status, no changes will be applied in the perioperative processes of our study patients.

Epworth sleepiness score questionnaire (Epworth Sleepness score), SF-12 quality of life questionnaire and STOP-BANG scores, mallampati score, cormack- lahane score, weight and neck circumference measurements will be taken again when the patients come to the control for surgery in the sixth postoperative month.

The changes of these values compared to preoperative values will be analysed at the sixth month after the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65
* American society of assosication score (ASA) :1-3
* To undergo Obstructive sleep apnea surgery (OSAS)

Exclusion Criteria:

* Verbal and written consent cannot be obtained

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years with American society of anaesthesiologist score 1-3 who will undergo obstructive sleep apnoea surgery
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Change of Modified mallampati score | post operative sixth month
  Modified mallampati score is one of the difficult airway markers evaluated preoperatively When the mouth is opened and the tongue is protruded Grade 1:soft palate, uvula, plicae and tonsils are clearly visible Grade 2:The soft palate, uvula, plicae and upper pole of the tonsils are visible.
  Grade 3: only the soft palate and part of the palate can be seen. Grade 4:only the hard palate can be seen.

SECONDARY OUTCOMES:
Sleep quality assesment pre and post operative surgery | post operative sixth month
  Eppworth sleepiness test (ESS) The ESS subjectively measures sleepiness as it occurs in ordinary life situations.It can be used to screen for excessive sleepiness or to follow an individual's subjective response to an intervention.
  Eight situations are described on a questionnaire:
  * Sitting and reading
  * Watching television
  * Sitting inactively in a public place
  * Riding as a passenger in a car for one hour without a break
  * Lying down to rest in the afternoon when circumstances permit
  * Sitting and talking with someone
  * Sitting quietly after lunch without alcohol
  * Sitting in a car as the driver, while stopped for a few minutes in trafficEach situation receives a score of 0 to 3, which is related to the likelihood that sleep will be induced:
  * 0 = would never doze
  * 1 = slight chance of dozing
  * 2 = moderate chance of dozing
  * 3 = high chance of dozing
  Total ESS score can range from 0 to 24, with higher scores correlating with increasing degrees of sleepiness
Change of Cormack lahane score | post operative sixth month
  Cor Mack Lahane Score:The Cormack-Lehane scale describes the best view of the glottis during laryngoscopy, with grades defined by the structures that can be seen, as follows:
  Grade 1 - Most of the glottis Grade 2 - Only the posterior extremity of the glottis Grade 3 - Only the epiglottis Grade 4 - Neither the glottis nor the epiglottis

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Sencan, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmıt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing of patient data is prohibited by the organisation. If necessary, it can be accessed by obtaining the relevant permissions

REFERENCES:
- [Background] Koh W, Kim H, Kim K, Ro YJ, Yang HS. Encountering unexpected difficult airway: relationship with the intubation difficulty scale. Korean J Anesthesiol. 2016 Jun;69(3):244-9. doi: 10.4097/kjae.2016.69.3.244. Epub 2016 Jun 1. PMID 27274369
- [Background] Kollmeier BR, Boyette LC, Beecham GB, Desai NM, Khetarpal S. Difficult Airway. 2023 Apr 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470224/ PMID 29261859
- [Background] Mark LJ, Herzer KR, Cover R, Pandian V, Bhatti NI, Berkow LC, Haut ER, Hillel AT, Miller CR, Feller-Kopman DJ, Schiavi AJ, Xie YJ, Lim C, Holzmueller C, Ahmad M, Thomas P, Flint PW, Mirski MA. Difficult airway response team: a novel quality improvement program for managing hospital-wide airway emergencies. Anesth Analg. 2015 Jul;121(1):127-139. doi: 10.1213/ANE.0000000000000691. PMID 26086513